CLINICAL TRIAL: NCT00891124
Title: A Multi-center, Prospective, Observational Study to Assess the Effect of Patient Education Related to CV Risk Factors in Type 2 Diabetes Mellitus
Brief Title: Effect of PATient Education Related to CV Risk factOrs in Type 2 Diabetes Mellitus(Patrol).
Acronym: PATROL
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: AstraZeneca, AstraZeneca
Other Study IDs: NIS-CKR-DUM-2009/2
Record Dates: First submitted 2009-04-28; First posted 2009-05-01 (Estimated); Last update posted 2009-11-03 (Estimated); Status verified 2009-11

CONDITIONS: Glycemia; Hypertension; Hyperlipidemia
Keywords: Hypertension; Type II DM; Hyperlipidemia; Glycemia; ADA 2008 guideline; Patient Consultation
MeSH Terms: conditions — Hypertension; Hyperlipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Type II DM and Hypertension and/or Hyperlipidemia

SUMMARY:
This study will address the proportion of achievement patients in treatment target goal on glycemic control, hypertension and hyperlipidemia according to ADA 2008 guideline, among outpatients coming to the Korean primary care nationwide.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had been diagnosed with type II diabetes mellitus
* Patients with hypertension and / or hyperlipidemia
* Patients who had agreed to Informed

Exclusion Criteria:

* Patients who had been diagnosed with type I diabetes mellitus
* Patients with neither hypertension and hyperlipidemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type II DM and Hypertension and/or Hyperlipidemia
Sampling Method: Non-Probability Sample
Enrollment: 4045 (Actual)
Dates: Start 2009-05; Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Proportion of achievement patients in treatment target goal on glycemic control, hypertension and hyperlipidemia according to ADA 2008 guideline | At baseline and Endpiont (after 2months)

SECONDARY OUTCOMES:
The treatment goal of risk factors is based on ADA guideline. | At baseline and Endpiont (after 2months)

CONTACTS AND LOCATIONS:
Overall Officials: Joonwoo Bahn, Study Director — ASTRAZENECA, Korea Medical Department
Locations (7):
- South Korea (7):
  - Research Site, Busan
  - Research Site, Cheiju
  - Research SIte, Daegu
  - Research Site, Gwangju
  - Research Site, Hongseong
  - Research Site, Seoul
  - Research Site, Sungman